CLINICAL TRIAL: NCT02198235
Title: Prolonged Popliteal Fossa Nerve Blockade
Brief Title: Prolonged Popliteal Fossa Nerve Blockade (Prolonged Pop)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2012-017
Record Dates: First submitted 2012-09-21; First posted 2014-07-23 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control NB + IV Dex + IV Bup (Active Comparator): IV Dexamethasone (4 mg) + IV Buprenorphine (150 mcg)
  Interventions: Drug: Dexamethasone; Drug: Buprenorphine
- Control NB + IV Dex (Active Comparator): IV Dexamethasone (4 mg)
  Interventions: Drug: Dexamethasone
- NB with Dex + Bup in block. (Experimental): Dexamethasone (4 mg) Buprenorphine (150 mcg)
  Interventions: Drug: Dexamethasone; Drug: Buprenorphine

INTERVENTIONS:
Drug: Dexamethasone
Drug: Buprenorphine
  Arms: Control NB + IV Dex + IV Bup; NB with Dex + Bup in block.

SUMMARY:
This study looks at addition of medications to the local anesthetic for the nerve blockade.

DETAILED DESCRIPTION:
Following major foot and ankle surgery patients complain of severe pain. Currently, Hospital for Special Surgery (HSS) usually uses nerve blocks (injections of local anesthetic near nerves supplying the lower leg) to help manage pain after this type of surgery. Patients also receive additional pain pills, including narcotics as needed. This study looks at addition of medications to the local anesthetic for the nerve blockade. The investigators hope that these medications (dexamethasone and buprenorphine) will prolong the pain relief from the nerve block. There are 3 groups in the study. One group is a control, and receives usual therapy: nerve block + pain pills. This is typically what the patient would receive as standard care if they were not in the study. One group uses a nerve block with additives (+ pain pills). One group gets a nerve block (local anesthetic only) + pain pills + intravenous buprenorphine - this is meant to see if the buprenorphine acts directly on the nerve that was blocked, or indirectly acts on the brain.

Patients will be followed while in the hospital, and contacted by telephone and/or email after discharge for 2-3 days. Patients will be asked about their pain levels and the duration of their block. The investigators will enroll 90 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Dr. Levine or Dr. Roberts at Hospital for Special Surgery
* Patients aged 18-75
* Patients scheduled for discharge from HSS after foot or ankle surgery
* A single-injection popliteal fossa nerve block is judged appropriate
* Surgery confined to foot and ankle (no iliac crest bone graft planned - iliac aspirate is not an exclusion criterion)

Exclusion Criteria:

* < 18 and > 75
* Surgery that will cause pain at sites outside the distal lower extremity (e.g. iliac crest bone graft)
* Bilateral surgery
* Chronic pain (defined as regular use of opioid analgesics for > 3 months)
* Chronic use of steroids (defined as regular use of steroids for > 3 months)
* Contraindication to performance of the popliteal fossa nerve block with 30 cc 0.25% bupivacaine (e.g. alleged bupivacaine sensitivity, low body weight, etc.)
* Contraindications to dexamethasone or buprenorphine (e.g. allergy, insulin dependent diabetes mellitus, etc.)
* Patients who have been diagnosed with altered pain perception or have lack of sensation
* Inability of the patient to describe postoperative pain (e.g. psychiatric disorder, dementia)
* Non-English speaking patients (the questionnaire is in English, and translations would have to be separately validated)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital For Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] YaDeau JT, Paroli L, Fields KG, Kahn RL, LaSala VR, Jules-Elysee KM, Kim DH, Haskins SC, Hedden J, Goon A, Roberts MM, Levine DS. Addition of Dexamethasone and Buprenorphine to Bupivacaine Sciatic Nerve Block: A Randomized Controlled Trial. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):321-9. doi: 10.1097/AAP.0000000000000254. PMID 25974277

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Nerve Block + IV Dexamethasone: IV Dexamethasone (4 mg)
  Dexamethasone
- Control Nerve Block + IV Dexamethasone + IV Buprenorphine: IV Dexamethasone (4 mg) + IV Buprenorphine (150 mcg)
  Dexamethasone
  Buprenorphine
- Nerve Block With Dexamethasone + Buprenorphine in Block.: Dexamethasone (4 mg) Buprenorphine (150 mcg)
  Dexamethasone
  Buprenorphine
Period: Overall Study
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Started | 30 | 30 | 30
Completed | 27 | 28 | 28
Not Completed | 3 | 2 | 2
Not completed — Lost to Follow-up | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block. | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (15.9) | 51.1 (15.3) | 52.8 (14.2) | 51.7 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 17 | 51
  Male | 14 | 12 | 13 | 39
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (5.68) | 26.3 (4.37) | 26.3 (5.16) | 26.6 (5.05)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Score With Movement
Description: Pain with movement at 24 hours from the nerve block (0-10; 0 = no pain, 10 = worst possible pain)
Time Frame: 24 hours after the popliteal block is given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Number analyzed (Participants) | 27 | 28 | 28
units on a scale | 1.9 (2.6) | 1 (1.6) | 1.3 (2.1)

2. Secondary Outcome: Block Duration
Description: When did the nerve block entirely wear off?
Time Frame: 24 hours and 48 hours after the popliteal block is given
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Number analyzed (Participants) | 27 | 28 | 28
hours | 30 [24.1 to 45.2] | 37.9 [30.7 to 43.9] | 45.6 [33.9 to 53.8]

3. Secondary Outcome: Numeric Rating Scale (NRS) Pain Score at Rest
Description: Pain at rest at 24 hours from the nerve block (0-10; 0 = no pain, 10 = worst possible pain)
Time Frame: 24 hours after the popliteal block is given
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Number analyzed (Participants) | 27 | 28 | 28
units on a scale | 1.8 (2.5) | .9 (1.3) | .8 (1.6)

4. Secondary Outcome: Median Time to Requiring Oral Opioids
Description: Did patient have pain requiring oral opioids?
Time Frame: 24 hours after the popliteal block is given
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Number analyzed (Participants) | 27 | 28 | 28
hours | 25.5 [18.0 to 34.7] | 30 [26.8 to 40.5] | 35.3 [30.3 to 55.8]

ADVERSE EVENTS:
Arm/Group | Control Nerve Block + IV Dexamethasone | Control Nerve Block + IV Dexamethasone + IV Buprenorphine | Nerve Block With Dexamethasone + Buprenorphine in Block.
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes